CLINICAL TRIAL: NCT06887192
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of ML-007C-MA for the Treatment of Hallucinations and Delusions Associated With Alzheimer's Disease Psychosis
Brief Title: A Study to Assess the Efficacy and Safety of ML-007C-MA for the Treatment of Alzheimer's Disease Psychosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MapLight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ML-007C-MA-221; 2024-519820-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-05

CONDITIONS: Psychosis Associated With Alzheimer's Disease
Keywords: Alzheimer Disease; Brain Diseases; Central Nervous System Diseases; Delusions; Dementia; Hallucinations; Mental Disorders; Nervous System Diseases; Neurocognitive Disorders; Neurodegenerative Diseases; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Tauopathies
MeSH Terms: conditions — Alzheimer Disease; Brain Diseases; Central Nervous System Diseases; Delusions; Dementia; Hallucinations; Mental Disorders; Nervous System Diseases; Neurocognitive Disorders; Neurodegenerative Diseases; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Tauopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ML-007C-MA (Experimental)
  Interventions: Drug: ML-007C-MA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ML-007C-MA — ML-007C-MA dosed as 105/1.5 mg (one tablet of 105/1.5 mg ML-007C-MA), or 210/3 mg (two tablets of 105/1.5 mg ML-007C-MA )
  Arms: ML-007C-MA
Drug: Placebo — Placebo Tablets
  Arms: Placebo

SUMMARY:
ML-007C-MA-221 is a Phase 2, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of ML-007C-MA in male and female participants aged 55 to 90 years with hallucinations and delusions associated with Alzheimer's Disease Psychosis (ADP).

The primary objective is to evaluate the efficacy of ML-007C-MA compared with placebo for the treatment of hallucinations and delusions associated with ADP as measured by the Neuropsychiatric Inventory-Clinician (NPI-C): Hallucinations and Delusions (H+D) score.

ELIGIBILITY:
Key Inclusion Criteria:

1. Willing and able to provide written informed consent, or, if deemed lacking in the capacity to provide informed consent, the following requirements for consent must be met:

   1. The participant's LAR (or care partner, if local regulations allow) must provide written informed consent AND
   2. The participant will provide written (if capable) informed assent.
2. Aged 55 to 90 years, inclusive, at time of informed consent.
3. Meets clinical criteria for Possible AD or Probable AD.
4. Presence of psychotic symptoms (meeting International Psychogeriatric Association criteria) (Cummings 2020) for at least 2 months before Screening.
5. Has resided at the same home, residential assisted living, or nursing home facility for a minimum of 6 weeks before Screening.
6. Has a designated care partner who is in contact with the participant frequently enough to accurately report on the participant's symptoms and adherence to study drug.
7. Has a NPI-C H+D score of ≥ 6 AND meet at least 1 of the following criteria:

   1. Moderate to severe delusions, defined as NPI-C Delusions domain score of ≥ 2 on at least 2 of the 8 items OR
   2. Moderate to severe hallucinations, defined as NPI-C Hallucinations domain score of ≥ 2 on at least 2 of the 7 items.
8. Has a (CGI)-S hallucinations and delusions domain-specific score ≥4
9. Has an Mini-mental State Examination (MMSE) score of 6 to 26, inclusive.

Key Exclusion Criteria:

1. Under the care of hospice, bed-bound, or receiving end-of-life palliative care.
2. Psychotic symptoms that are primarily attributable to substance abuse or a medical, neurological or psychiatric condition other than Alzheimer's disease.
3. Evidence of a CNS disorder other than Alzheimer's disease that is the primary cause of, or a significant contributor to the participant's dementia.
4. Moderate or severe major depressive episode within 3 months of Screening, according to DSM-5 criteria.
5. Has had an amyloid positron emission tomography (PET) brain scan or cerebrospinal fluid (CSF) Alzheimer's disease biomarker test in the past 3 years with results inconsistent with a diagnosis of AD.
6. Evidence of a clinically significant and/or unstable medical condition that, in the opinion of the investigator or medical monitor, could substantially impair cognition, compromise participant safety, interfere with the participant's ability to comply with study procedures or substantially impair the evaluation of efficacy or safety assessments.
7. Gastric retention, urinary retention or narrow-angle (angle-closure) glaucoma
8. Meets or has met DSM-5 criteria for alcohol or substance use disorder within the past 12 months (excluding caffeine and nicotine).
9. Has previously participated in any clinical study with ML-007 or ML-007C-MA.
10. Received or may have received an investigational drug, biological product or device within 90 days before Baseline (or 6 months for investigational Alzheimer's disease-modifying therapies).

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to End of Treatment in the Neuropsychiatric Inventory-Clinician: Hallucinations and Delusions (NPI-C H+D) score | Baseline and End of Treatment (7 weeks)
  NPI-C H+D scale includes 2 domains from the NPI-C scale, namely, hallucinations and delusions. These 2 domains include the following number of items to be rated by the clinician: Hallucinations, 7 items (maximum score = 21) and Delusions, 8 items (maximum score = 24). The maximum score for the NPI-C: H+D scale is 45. Higher scores on this scale indicate worse outcomes.

SECONDARY OUTCOMES:
Change from Baseline to End of Treatment in the Clinical Global Impressions-Severity (CGI-S) hallucinations and delusions domain-specific score | Baseline and End of Treatment (7 weeks)
  The CGI-S scale is a clinician-rated, 7-point scale that is designed to rate the severity of the participant's hallucinations and delusions using the investigator's judgment and past experience with participants who have Alzheimer's disease psychosis. Higher scores on this scale indicate worse outcomes.
Change from Baseline to End of Treatment in the Neuropsychiatric Inventory - Clinician Agitation and Aggression (NPI-C A+A) score in participants who have a CGI-S agitation/aggression domain-specific score of ≥4 at Baseline | Baseline and End of Treatment (7 weeks)
  NPI-C A+A scale includes 2 domains from the NPI-C scale, namely, agitation and aggression. These 2 domains include the following number of items to be rated by the clinician: Agitation, 13 items (maximum score = 39), and Aggression, 8 items (maximum score = 24). The maximum score for the NPI-C A+A scale is 63. Higher scores on this scale indicate more severe symptoms of agitation and aggression.

CONTACTS AND LOCATIONS:
Overall Officials: MapLight Therapeutics, Study Director — MapLight Therapeutics
Locations (20):
- United States (16):
  - Clinical Site, Scottsdale, Arizona
  - Clinical Site, Tucson, Arizona
  - Clinical Site, Anaheim, California
  - Clinical Site, Orange, California
  - Clinical Site, Boca Raton, Florida
  - Clinical Site, Deerfield Beach, Florida
  - Clinical Site, Doral, Florida
  - Clinical Site, Homestead, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Miami Gardens, Florida
  - Clinical Site, Naples, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, West Palm Beach, Florida
  - Clinical Site, Las Vegas, Nevada
  - Clinical Site, West Long Branch, New Jersey
  - Clinical Site, Independence, Ohio
- Canada (4):
  - Clinical Site, Brampton, Ontario
  - Clinical Site, London, Ontario
  - Clinical Site, Toronto, Ontario
  - Clinical Site, Lévis, Quebec

IPD SHARING:
Plan to Share IPD: No